CLINICAL TRIAL: NCT05315245
Title: Acute Gastrointestinal Injury in Critically Ill Children in Pediatric Intensive Care Unit of Cipto Mangunkusumo Hospital
Brief Title: Acute Gastrointestinal Injury in Pediatrics
Acronym: AGI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Antonius Hocky Pudjiadi, SpA(K), Principal Investigator, Indonesia University
Other Study IDs: 19-04-0471
Record Dates: First submitted 2020-09-18; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Acute Gastrointestinal Injury; Gastrointestinal Failure; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AGI — no intervention, only observation

SUMMARY:
Critically Ill children may develop acute gastrointestinal injury secondary to severe inflammation.

DETAILED DESCRIPTION:
Data collection from enrolled subjects including profile, laboratory examinations, inflammatory markers on day 1 and day 3, nutritional support and daily calorie intake, and finally outcome of the patient

ELIGIBILITY:
Inclusion Criteria:

* critically ill pediatric patients receiving care at the PICU
* presence of AGI (any degree)

Exclusion Criteria:

* patients who's body weight cannot be measured

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All critically ill patients admitted to PICU
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
PELOD-2 score | time of AGI diagnosis, day-1 PELOD-2 score
  The Pediatric Logistic Organ Dysfunction (PELOD)-2 score is used to predict mortality and assess organ dysfunction. It consist of 10 components, assessing 5 organ dysfunction. The minimum score of PELOD-2 is 0 and the maximum score is 33. With the increasing organ dysfunction, the probability of death also increases.
mortality | days from PICU admission date up to 28 days follow-up
  PICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Antonius H Pudjiadi, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided